CLINICAL TRIAL: NCT00223197
Title: A Double-blind Placebo Controlled Trial of Pregnenolone for Depression in Patients With Bipolar Disorders or Recurrent Major Depressive Disorder and a History of Substance Abuse
Brief Title: Pregnenolone Trial for Depression in Bipolar Disorders or Recurrent Major Depressive Disorder With Substance Abuse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1103-714
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2006-08

CONDITIONS: Bipolar Disorder; Major Depressive Disorder; Substance Abuse
Keywords: Bipolar with depression; Recurrent major depressive disorder; substance abuse dependence
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Substance-Related Disorders | interventions — Pregnenolone

INTERVENTIONS:
Drug: Pregnenolone

SUMMARY:
The purpose of this research is to determine if pregnenolone supplement is associated with a reduction in substance use and craving in patients with recurrent major depressive disorder or bipolar disorder and substance abuse/dependence. This research also wants to explore if pregnenolone supplements are associated with improvement in psychiatric symptoms and memory, which are often negatively affected in these patients. It is hypothesized that patients receiving pregnenolone supplements would show greater improvements in mood symptoms and memory, and crave substances less than the patients receiving placebo.

DETAILED DESCRIPTION:
Seventy five - (75) outpatients meeting the inclusion and exclusion criteria will be enrolled after completing an IRB-approved informed consent process. Baseline evaluation will include a medical and psychiatric history, structured clinical interview for DSM-IV (SCID), mood assessment with the Hamilton Rating Scale for Depression (HRSD, 17-item version), Inventory of Depressive Symptomatology-Self Report (IDS-SR) (Rush et al., 1996), Hamilton Rating Scale for Anxiety (HRSA), Young Mania Rating Scale (YMRS), and, and cognitive assessment with the Rey Auditory Verbal Learning Test (RAVLT), Stroop Test Color Trails, Wechsler Test of Adult Reading and the Brief Visual Memory Test-Revised (BVMT-R) will be performed. Substance use (days/week) of use, urine drug screens and time to relapse will be monitored. Craving for substances will be monitored with visual analogue scales. Pregnenolone or placebo will be initiated at one capsule/day (50 mg/d if active medication). Pregnenolone and the placebo will be obtained from Abrams Pharmacy, which has ensured the potency (the supplier uses GMP pharmaceutical standards). Participants will return for reassessment every 2 weeks for 8 weeks with the HRSD, IDS-SR, YMRS, ISS, and a neurocognitive battery (e.g. RAVLT, Stroop Test and Trails B). Side effects will be monitored with the PRD-III Somatic Symptom Scale (Thase et al., 1996). At week 4 subjects who not having significant side effects and have not had a 50% reduction in HRSD scores will have the dosage increased to two capsules per day (100 mg/d if active medication). Participants will be paid $30 at weeks 2, 4, and 8. Participants who respond favorably will, at completion, have the option of continuing this over-the-counter supplement if they so choose with their physician's knowledge and approval.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of Bipolar I, II, NOS or recurrent major depressive disorder
* Bipolar I patients must be receiving a mood stabilizer
* History of substance-related disorder with no substance use within 14 days of beginning the study

Exclusion Criteria:

* Currently suicidal or homicidal (within 4 weeks of study enrollment)
* Severe or life-threatening medical illness
* Pregnant or nursing female
* Current pregnenolone therapy or allergies to pregnenolone
* Member of vulnerable population (prisoner, demented, mental retardation)
* Participants with treatment resistant depression
* Actively psychotic within 2 months prior to enrollment;
* A change in antipsychotic medication 1 month prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2004-02; Study Completion 2006-04

PRIMARY OUTCOMES:
For the primary outcome measure, we will analyze both between group differences in change from baseline but also response rates.
Paired T tests will be used to compare outcome measures of HRSD, IDS-SR, HRSA, YMRS, RAVLT, Stroop, Trails B, and PRD III from baseline to exit.
All participants returning for at least one post baseline assessment will be used.
In the case of early withdrawal from the study, the last visit will be used for the exit scores (last observation carried forward).

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, M.D., Ph.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States